CLINICAL TRIAL: NCT05294978
Title: Qualification for Cone-Optogenetics (EyeConic)
Brief Title: EyeConic: Qualification for Cone-Optogenetics
Status: Recruiting | Type: Observational
Sponsor: Institute of Molecular and Clinical Ophthalmology Basel (Other)
Responsible Party: Sponsor
Other Study IDs: IOB_EyeConic_2021
Record Dates: First submitted 2022-02-16; First posted 2022-03-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Retinal Dystrophies
Keywords: Cone-Optogenetics; Rod-cone Dystrophy; Cone-rod Dystrophy; Generalized retinal dystrophies; Inherited retinal disease
MeSH Terms: conditions — Retinal Dystrophies; Cone-Rod Dystrophies | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: -Availability of macular optical coherence tomography (OCT)
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)
- Controls: -Availability of macular optical coherence tomography (OCT)
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography (OCT) — Data of macular optical coherence tomography (OCT)

SUMMARY:
This study aims to prepare for the first-in-human clinical trial of cone optogenetics vision restoration. As a first step, this worldwide multicenter ocular imaging study (EyeConic Study) is performed to identify eligible patients.

DETAILED DESCRIPTION:
In a subset of patients with inherited retinal dystrophies (IRDs), cones lose their light-sensitive outer segments but remain alive in a dormant stage. This creates an opportunity to resensitize them through targeted optogenetic tools. However, the true proportion of low vision patients harboring dormant, non-functional cones, is currently unknown. The worldwide multicenter retrospective study (EyeConic) aims to estimate the proportion of low vision patients with remaining cone cell bodies for the first time.

ELIGIBILITY:
Inclusion Criteria (patients):

* Diagnosis of generalized IRD
* Low vision as defined as visual acuity worse or equal to 0.05 (or 20/400) in the study eye
* Availability of macular optical coherence tomography (OCT)

Inclusion Criteria (controls):

* Normal ophthalmic findings
* Availability of macular optical coherence tomography (OCT)

Exclusion Criteria (all):

* Other eye diseases with a significant effect on vision or retinal structure
* Extraocular disease affecting retinal structure such as neurodegenerative diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with diagnosis of generalized retinal dystrophy
  * Normal controls
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
OCT - Central retinal volume | Baseline (about 10 minutes)
  Number of participants with preserved central retinal volume

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Feltgen, MD, Principal Investigator — University Hospital Basel/Institute of Molecular and Clinical Ophthalmology Basel, Switzerland
Locations (9):
- United States (3):
  - University of California San Francisco, Department of Ophthalmology, San Francisco, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - University of Pittsburgh, Department of Ophthalmology, Pittsburgh, Pennsylvania
- Beijing Institute of Ophthalmology, Beijing, China
- Universitätsklinikum Tübingen Augenklinik, Tübingen, Germany
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary
- Oculista Ospedale Parma, Parma, Italy
- University Hospital Basel, Eye Clinic, Basel, Switzerland
- Moorfields Eye Hospital, London, United Kingdom